CLINICAL TRIAL: NCT02612597
Title: The Effect of Blood Volume Changes After Bed Rest and Aerobic Exercise Training on the Glucose Tolerance
Brief Title: The Effect of Blood Volume Changes on the Glucose Tolerance
Acronym: BV-GT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carsten Lundby (Other)
Responsible Party: Sponsor-Investigator, Carsten Lundby, Prof. Dr., Zurich Center for Integrative Human Physiology
Organization: Zurich Center for Integrative Human Physiology (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-Nr. 2015-0453
Record Dates: First submitted 2015-11-13; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Healthy; Overweight
Keywords: before and after bedrest; healthy untrained; before and after exercise training
MeSH Terms: conditions — Overweight | interventions — Bed Rest; Exercise

ARMS (2):
- Bedrest (Experimental): 4 days of bedrest
  Interventions: Other: Bedrest
- Exercise Training (Experimental): 6 weeks of aerobic endurance exercise training with 4 supervised sessions per week at an average intensity of 65 % of maximal heart rate
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Bedrest
  Arms: Bedrest
Other: Exercise Training
  Arms: Exercise Training

SUMMARY:
In this study the investigators would like to elaborate on the mechanisms that lead to a higher insulin sensitivity after exercise training and a lower insulin sensitivity after bedrest.

The investigators speculate that the concomitant chances in blood volume during training and bedrest might explain the changed insulin sensitivity because with a changing blood volume also the dilution space of the glucose will change.

Furthermore, the investigators would like to work on the influence of a changed capacity of skeletal muscle for glucose uptake and glycogen storage on the glucose sensitivity.

Therefore, A) a bed rest study with healthy untrained subjects and B) a training study with obese pre-diabetic patients will be conducted.

DETAILED DESCRIPTION:
While there is little doubt that physical inactivity leads to reduced insulin sensitivity and in contrast hereto that physical activity improves insulin sensitivity the underlying mechanisms are still to a large extend unknown. With this study the investigators wish to test two independent hypotheses that may explain the observed changes:

The first hypothesis is that part of the explanation for the known increase in circulating levels of glucose in response to an oral glucose tolerance test (indicating reduced insulin sensitivity) following bed rest is due to a concomitantly reduced blood volume and thereby dilution space.

In addition the investigators also speculate that the reduced glucose response to an oral glucose tolerance test (indicating improved insulin sensitivity) after a training period is related to the exercise induced increase in blood volume, and hence an increased dilution space.

Based on this, the hypothesis to be tested with these two experimental approaches (bed rest and aerobic exercise training), is that at least part of the changes observed in the glucose tolerance following bed rest and aerobic exercise training are related to concomitantly occurring changes in blood volume.

The second hypothesis to be tested is that another important contributor to the changes in circulating glucose levels following an oral glucose tolerance test after bed rest and physical training are related to diminished or improved capacity for skeletal muscle glucose uptake and glycogen storage, respectively. The rationale here fore are that exercise training increases skeletal muscle glycogen content and storage capacity in healthy and type 2 diabetic patients, respectively, and that bed rest does the opposite.

To test this hypothesis two different intervention studies will be conducted. Study 1 is a bed rest study with healthy untrained subjects and study 2 is a training study with obese "pre-diabetic patients".

ELIGIBILITY:
Bedrest:

Inclusion Criteria:

* Informed consent as documented by signature
* Age: 18-35
* healthy (no chronic diseases)
* BMI: 19-25
* maximal oxygen uptake: 35-50 ml O2/min/kg

Exclusion Criteria:

* chronic diseases
* any health problems that do not allow the subjects to participate in the measurements (i.e. heart defect)
* History of familiar history (1st grade relatives) of venous thrombic-embolism or renal insufficiency
* Blood donation in the last month
* Any medication with known influence on blood volume, glucose metabolism and body weight
* Stay above 2500 m for more than 1 day
* Known allergies against Fragmin or Heparin

Training:

Inclusion criteria:

* Informed consent as documented by signature
* Age: 35-50
* BMI: 30-40
* Fat%: 30-40 %
* maximal oxygen uptake: 20-35 ml O2/min/kg
* HbA1c: 5.5 - 7.0 %

Exclusion criteria:

* Chronic diseases
* Any health problems that do not allow the subjects to participate in the measurements (i.e. heart defect)
* Blood donation in the last month
* Any medication with known influence on blood volume, glucose metabolism and body weight
* Stay above 2500 m for more than 1 day

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change in blood volume | Baseline and 4 days
Change in glucose tolerance | Baseline and 4 days
Change in blood volume | Baseline and 6 weeks
Change in glucose tolerance | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Lundby, Prof. Dr., Principal Investigator — Institute of Physiology, University of Zurich
Locations (1):
- Institute of Physiology, University of Zurich, Zurich, Canton of Zurich, Switzerland